CLINICAL TRIAL: NCT00148629
Title: Preventing Unnecessary Blood Transfusions in Pregnant Women in Africa Through Effective Primary Health Care
Brief Title: Treatment and Prevention of Severe Anemia in Pregnant Zanzibari Women
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cornell University (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); UNICEF (Other); Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: UCHS 02-10-030
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: Anemia; Low Birth Weight; Neonatal Mortality
Keywords: Anemia; Birth weight; Neonatal Mortality; Tanzania; Pregnancy
MeSH Terms: conditions — Anemia; Birth Weight | interventions — Geritol; Mebendazole

INTERVENTIONS:
Drug: multivitamin, mebendazole

SUMMARY:
The purpose of this research is to compare the efficacy of two low-cost low intervention packages to prevent and treat severe anemia in pregnant women in Zanzibar, Tanzania. The two packages are Standard of Care as described by the WHO (presumptive treatment for malaria and helminths plus daily iron + folic acid supplements) and Enhanced Care (Standard of Care plus daily multivitamins and a 2nd dose of anthelminthic.)

DETAILED DESCRIPTION:
This is a clinic-randomized trial involving 8 antenatal clinics and approximately 2500 women. The specific aims are:

Aim 1: To evaluate the efficacy of the current internationally recommended standard of care, as described by the WHO, for the prevention of severe anemia among pregnant Zanzibari women. This aim will be achieved through a pre-post intervention comparison.

Aim 2: To evaluate the efficacy of an enhanced treatment regimen in comparison to the current standard of care to prevent severe anemia among pregnant Zanzibari women.

Aim 3: To evaluate the efficacy of the current internationally recommended standard of care, as described by the WHO, for the cure of severe anemia among pregnant Zanzibari women.

Aim 4: To evaluate the efficacy of an enhanced treatment regimen in comparison to the current standard of care to cure severe anemia among pregnant Zanzibari women.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman

Exclusion Criteria:

* Not a permanent resident of the community

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2500
Dates: Start 2004-04

PRIMARY OUTCOMES:
Incidence of severe anemia (Hb < 7 g/dL)
Cure of severe anemia

SECONDARY OUTCOMES:
Infant birth weight
Neonatal mortality
Neonatal morbidity
Blood loss during delivery

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca J Stoltzfus, PhD, Principal Investigator — Cornell University; James M Tielsch, PhD, Principal Investigator — The Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Public Health Laboratory "Ivo de Carneri", Wawi, Zanzibar, Tanzania